CLINICAL TRIAL: NCT05629182
Title: Potential Injury Incidents At the FIFA World Cup Qatar 2022
Status: Completed | Type: Observational
Sponsor: Federation Internationale de Football Association (Other)
Responsible Party: Sponsor
Other Study IDs: 005
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention applied - Observational study only — Observational study only. Video footage is used to review all 64 matches in the football tournament.

SUMMARY:
This is an exploratory observational study.

Video footage is used to review all 64 matches in the football tournament.

All players actions are registered using the FIFA football language, such as, pass completed, clearance, etc.

Potential injury incidents are registered, and for each incident the injury location, contact type, player reaction, velocity, location, game reaction, referee reaction, medical staff on pitch, and outcome (e.g. substitution) are also registered.

DETAILED DESCRIPTION:
Video footage is used to review all 64 matches in the FIFA World Cup Qatar 2022.

All players actions are registered using the FIFA football language, such as, pass completed, clearance, etc.(https://www.fifatrainingcentre.com/en/resources-tools/football-language/index.php)

Potential injury incidents are registered, and for each incident the injury location, contact type, player reaction, velocity, location, game reaction, referee reaction, medical staff on pitch, and outcome (e.g. substitution) are also registered.

Simple descriptive statistics are used to create overviews of the outcomes described above, including comparisons between actions which do or do not lead to potential injury incidents.

A secondary analysis may be performed including injury diagnoses, if players consent as part of another study on injury surveillance allowing video analysis of their injuries.

No a priori sample size calculation was performed, as all potential injury incidents are included.

ELIGIBILITY:
Inclusion Criteria:

* All participating football players at the FIFA World Cup Qatar 2022.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The tournament includes 32 national teams, and each team is allowed to select 26 players, giving at total of 832 potential participants. In total, 64 matches will be played over 29 days.
Sampling Method: Non-Probability Sample
Enrollment: 832 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Potential injury incidents | November-December 2022
  Potential injury incidents, defined as "when a player stays down for more than 5 seconds or a player indicates they are injured to the referee, teammates, their coach, or medical staff.

SECONDARY OUTCOMES:
Injury inciting circumstances | November-December 2022
  All players actions are registered using the FIFA football language, such as, pass completed, clearance, etc. For each potential injury incident, the injury location, contact type, player reaction, velocity, location, game reaction, referee reaction, medical staff on pitch, and outcome (e.g. substitution) are also registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Fèdèration Internationale de Football Association, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided